CLINICAL TRIAL: NCT05846789
Title: A Pragmatic Phase II Trial of SOC Chemotherapy +/- Tocilizumab for Metastatic Triple Negative and ER-low Breast Cancers
Brief Title: SOC Chemotherapy +/- Tocilizumab for Triple Negative and ER-low Breast Cancers
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kathy Miller (Other)
Collaborators: Genentech, Inc. (Industry); Breast Cancer Research Foundation (Other); Susan G. Komen Breast Cancer Foundation (Other)
Responsible Party: Sponsor-Investigator, Kathy Miller, Ballvé-Lantero Professor of Medicine, Indiana University
Organization: Indiana University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTO-IUSCCC-0817
Record Dates: First submitted 2023-04-27; First posted 2023-05-06 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Breast Cancer; Triple Negative Breast Cancer; Estrogen-receptor-low Breast Cancer
Keywords: Breast Cancer; Phase II
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — tocilizumab

STUDY DESIGN:
Intervention Model Description: Patients are stratified by either Black or non-Black (race-based cohort) and are then randomized 1:1 to either the monotherapy or combination arm. This requires 42 patients (21 per treatment arm) in stage I for each race-based cohort. If the no. of response in experimental - no. of response in control is no greater than -1, the trial is early stopped at stage I for futility. Otherwise, additional 42 patients for each race-based cohort will be enrolled and randomized to the study in stage II for a total of 168 subjects across all 4 arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Black Monotherapy (Active Comparator)
  Interventions: Drug: SOC Chemotherapy
- Black Combination treatment (Experimental)
  Interventions: Drug: SOC Chemotherapy; Drug: Tocilizumab
- Non-Black Monotherapy (Active Comparator)
  Interventions: Drug: SOC Chemotherapy
- Non-Black Combination treatment (Experimental)
  Interventions: Drug: SOC Chemotherapy; Drug: Tocilizumab

INTERVENTIONS:
Drug: SOC Chemotherapy — SOC Chemotherapy will be given AUC 6 IV q3 weeks for a maximum of 9 infusions.
Drug: Tocilizumab — Tocilizimab 8 mg/ actual body weight in kg IV q4 weeks
  Arms: Black Combination treatment; Non-Black Combination treatment

SUMMARY:
This is a randomized Phase II study of standard of care (SOC) chemotherapy monotherapy vs. SOC chemotherapy combined with tocilizumab in in Black and non-Black patients with metastatic triple negative or ER low breast cancer.

DETAILED DESCRIPTION:
Randomized phase II using a two-stage Bayesian optimal phase II two-arm design (BOP2). Patients are randomized 1:1 to either the monotherapy or combination arms. This requires 42 patients (21 per treatment arm) in stage I for each race-based cohort. If the no. of response in experimental - no. of response in control is no greater than -1, the trial is early stopped at stage I for futility. Otherwise, additional 42 patients for each race-based cohort will be enrolled and randomized to the study in stage II.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years old at the time of informed consent
2. Ability to provide written informed consent and HIPAA authorization
3. Locally recurrent (not amenable to local therapy with curative intent) or metastatic breast cancer that is triple negative or ER-low (ER and PR ≤ 9% weak staining)
4. Received up to 2 prior therapies for metastatic disease

   1. Prior (neo)adjuvant therapy will be considered one line of therapy for metastatic disease in patients who recur while on or within 12 months of completion of (neo)adjuvant therapy.
   2. Participation in this protocol as either first, second and third-line therapy is allowed.
5. Planned standard of care chemotherapy based on NCCN guidelines.

   1. Single agent therapy is preferred but use of combination regimens considered SOC by NCCN is allowed.
   2. Chemotherapy delivered via a SOC antibody-drug conjugate is allowed but ADCs may not be used in combination with other agents.
6. Patients with tumors that are PD-L1+ (CPS > 10) must have had prior exposure to an immune checkpoint inhibitor in the metastatic setting.

   1. Patients who received (neo)adjuvant IO therapy and progress while on or within 12 months of completion of (neo)adjuvant IO therapy may participate without additional IO treatment.
   2. Patients with major contraindications to immune therapy, may participate without IO exposure regardless of PD-L1 status in the first line setting.
   3. PD-L1 status is not required for patients in the second line setting.
7. Measurable disease based on RECIST 1.1 criteria.
8. Disease amenable to and consent for study-specific biopsy NOTE: If no disease amenable to biopsy is present at the time of second biopsy, subjects may continue participation in the study and further study specific biopsies will not be required.
9. ECOG PS 0 or 1
10. Patients with treated, asymptomatic CNS disease may participate if the patient is > 4 weeks from completion of CNS therapy (radiation and/or surgery), is clinically stable at the time of study entry, and is receiving stable or decreasing dose of corticosteroids. Brain MRI or head CT is required at screening for patients with known brain metastases.
11. Adequate organ function as indicated by:

    1. Total bilirubin < ULN (except in patients with documented Gilbert's disease, who must have a total bilirubin < 3.0 mg/dL)
    2. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 5.0 x ULN
    3. Creatinine clearance of > 50 mL/min using the Cockcroft-Gault formula
    4. Absolute neutrophil count (ANC) > 1.2 K/mm3
    5. Platelets > 75 K/ mm3
    6. Hgb > 9.0 g/dL
12. Women of childbearing potential must have a negative pregnancy test within 14 days of protocol registration. Women are considered to have childbearing potential (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) unless they meet one of the following criteria:

    1. Has undergone a hysterectomy or bilateral oophorectomy; or
    2. Has been naturally amenorrheic for at least 24 consecutive months.
13. Women of childbearing potential and men must agree to use effective contraception throughout the study and for 6 months after the last study treatment.

NOTE: Acceptable methods of birth control include abstinence, partner with previous vasectomy, placement of an intrauterine device (IUD), condom with spermicidal foam/gel/film/cream/suppository, diaphragm or cervical vault cap, or hormonal birth control (pills or injections).

Exclusion Criteria:

1. Prior treatment with or known contraindication to treatment with tocilizumab or other IL-6/IL-6R targeted agent
2. Active infection requiring parenteral antibiotics
3. Concurrent use of methotrexate or systemic corticosteroids other than stable or decreasing doses for management of CNS involvement
4. Active or symptomatic CNS disease
5. Patients with HER2+ disease Note: HER2 will be considered positive if scored 3+ by immunohistochemistry (IHC) or 2+ by IHC associated with a fluorescence in situ hybridization (FISH) ratio of > 2.0 or > 6 total HER2 gene copies per cell.
6. Patients with active malignancy other than breast cancer. Patients with prior malignancies without recurrence after standard treatment will not be excluded
7. Radiation therapy within 2 weeks of registration
8. Hormone therapy within 2 weeks of registration
9. Planned treatment with Olaparib or other PARP inhibitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2024-07-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | through study completion (i.e. up to 2 years)
Efficacy of tocilizumab in Black and non-Black patients | through study completion (i.e. up to 2 years)
  efficacy defined as using the difference in difference approach across race based cohorts
Progression-free survival | through study completion (i.e. up to 2 years)

SECONDARY OUTCOMES:
Safety of SOC chemotherapy monotherapy compared to SOC chemotherapy combined with tocilizumab using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v 5.0 | through study completion (i.e. up to 2 years)
Evaluate the differences in inflammatory pathways between Black and non-Black patients | Baseline
  Tumor PZP, IL-6, and phosphoSTAT3
Evaluate the impact of Duffy genotype on efficacy in Black patients | Baseline
  Tumor PZP, IL-6, and phosphoSTAT3 between Duffy-null, Duffy-heterozygous, and Duffy-wild type

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Miller, MD, Principal Investigator — Indiana University
Locations (6):
- United States (6):
  - Emory University, Atlanta, Georgia
  - IU Health Joe and Shelly Schwarz Cancer Center, Carmel, Indiana
  - Indiana University Melvin and Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Duke University, Durham, North Carolina